CLINICAL TRIAL: NCT01426048
Title: Long-term Outcome of the TVT Procedure Without Preoperative Urodynamic Examination
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Turku University, Finland, Turku University, Finland
Other Study IDs: 118/180/2008
Record Dates: First submitted 2011-07-25; First posted 2011-08-30 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients operated on with the TVT
  Interventions: Other: Gynaecological examination and a supine stress test, questionnaires

INTERVENTIONS:
Other: Gynaecological examination and a supine stress test, questionnaires — Gynaecological examination and a supine stress test, questionnaires

SUMMARY:
A follow-up study of 191 patients operated on with the TVT procedure between January 1998 and May 2000 at the Department of Obstetrics and Gynecology in the Turku City Hospital. After a mean of 10.5 years patients were invited to a follow-up visit. Subjective outcome was evaluated with condition-specific and general quality of life and health questionnaires. Objective outcome was evaluated with gynaecological examination and a supine stress test. Objective cure was defined as a negative stress test and no need for a reoperation for SUI and subjective cure.

ELIGIBILITY:
Inclusion Criteria:

* 191 patients operated on with the TVT procedure between January 1998 and May 2000 at the Department of Obstetrics and Gynecology in the Turku City Hospital

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 191 female patients with genuine or recurrent stress urinary incontinence or mixed incontinence operated on with the TVT procedure at the mean of 10.5 years ago.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2008-11; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Objective outcome of the TVT operation | 13.5 years
  Objective outcome was measured with negative stress test and no need for reoperation for stress urinary incontinence during the follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku university hospital, Turku, Finland